CLINICAL TRIAL: NCT00025779
Title: Methylphenidate for Hyperactivity and Impulsiveness in Children and Adolescents With Pervasive Developmental Disorders
Brief Title: Methylphenidate in Children and Adolescents With Pervasive Developmental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: N01 MH70009; N01 MH80011; N01 MH70010; N01 MH70001; DSIR CT
Record Dates: First submitted 2001-10-23; First posted 2001-10-24 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2008-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Autistic Disorder; Pervasive Development Disorders
Keywords: Hyperactivity; Distractibility; Impulsiveness; Pervasive Development Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Child Development Disorders, Pervasive; Spasm; Impulsive Behavior | interventions — Methylphenidate; Guanfacine

INTERVENTIONS:
Drug: methylphenidate
Drug: guanfacine

SUMMARY:
This study will evaluate the efficacy and safety of methylphenidate for treating hyperactivity, impulsiveness, and distractibility in 60 children and adolescents with Pervasive Developmental Disorders (PDD). Methylphenidate (Ritalin)is approved by the Food and Drug Administration for the treatment of children and adolescents with Attention Deficit Hyperactivity Disorder (ADHD). Data supporting its safety and effectiveness in treating ADHD symptoms in PDD are limited. Children and adolescents who do not show a positive response to methylphenidate will be invited to participate in a pilot study of the non-stimulant medication guanfacine (Tenex).

DETAILED DESCRIPTION:
The safety and efficacy of methylphenidate (MPH) in 60 children and adolescents with PDD and behavioral difficulties (such as hyperactivity, impulsiveness and distractibility) will be evaluated in a multi-dose, 4-week randomized, crossover, placebo-controlled study. The MPH study has three parts: a Test-Dose Period, a Double-Blind trial and an 8-Week Extension Period (open-label). After a screening visit, eligible children will start a 1-week Test-Dose Period. During this week, each child will be given the three MPH doses that are used in the Double-Blind trial to make sure there are no serious side effects. If problems are encountered at the high dose level, that dose will not be given in the Double-Blind phase. The Double-Blind phase lasts 4 weeks and consists of three different MPH dose levels and a week of placebo. Each treatment/dose is given for 1 week, and neither the researcher nor the participants' families will know whether the medication is placebo or MPH. Children who do well during this phase will continue on the best dose of MPH (determined during the Double-Blind phase) for an additional eight weeks (open-label).

Those who do not show significant improvement during the Double-Blind phase, do not tolerate MPH during the Test Dose Period, or are not able to take MPH before beginning the study are offered open-label treatment with guanfacine for 8 weeks.

Prior to randomization in the MPH trial OR entry into the open-label guanfacine trial, there will be a medication-free period for children who are currently on medication. The withdrawal will be conducted in clinically appropriate way (depending on drug and duration of treatment) to minimize withdrawal effects. This period is to establish a drug-free baseline measurement and to minimize drug-drug interaction. No participant will be withdrawn from a currently effective medication.

ELIGIBILITY:
* Diagnosis of PDD (including Asperger's Disorder and Autistic Disorder)
* Clinically significant symptoms of ADHD
* Mental age of at least 18 months
* Blood pressure within normal ranges for age and gender
* Weight 16 kg or more
* Absence of chronic tic disorder
* Absence of any medical condition that would be incompatible with the study treatments
* Absence of evidence of hypersensitivity to study treatments

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2001-10; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
hyperactivity, impulsiveness, and distractibility

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Arnold, MD, Study Chair — Ohio State University; Larry Scahill, Ph.D — Yale University
Locations (5):
- United States (5):
  - UCLA Neuropsychiatric Institute, Los Angeles, California
  - Yale Child Study Center, New Haven, Connecticut
  - Indiana University-Riley Hospital for Children, Indianapolis, Indiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Scahill L, McDougle CJ, Williams SK, Dimitropoulos A, Aman MG, McCracken JT, Tierney E, Arnold LE, Cronin P, Grados M, Ghuman J, Koenig K, Lam KS, McGough J, Posey DJ, Ritz L, Swiezy NB, Vitiello B; Research Units on Pediatric Psychopharmacology Autism Network. Children's Yale-Brown Obsessive Compulsive Scale modified for pervasive developmental disorders. J Am Acad Child Adolesc Psychiatry. 2006 Sep;45(9):1114-23. doi: 10.1097/01.chi.0000220854.79144.e7. PMID 16926619
- [Background] Scahill L, Aman MG, McDougle CJ, McCracken JT, Tierney E, Dziura J, Arnold LE, Posey D, Young C, Shah B, Ghuman J, Ritz L, Vitiello B. A prospective open trial of guanfacine in children with pervasive developmental disorders. J Child Adolesc Psychopharmacol. 2006 Oct;16(5):589-98. doi: 10.1089/cap.2006.16.589. PMID 17069547
- [Background] Posey DJ, Aman MG, McCracken JT, Scahill L, Tierney E, Arnold LE, Vitiello B, Chuang SZ, Davies M, Ramadan Y, Witwer AN, Swiezy NB, Cronin P, Shah B, Carroll DH, Young C, Wheeler C, McDougle CJ. Positive effects of methylphenidate on inattention and hyperactivity in pervasive developmental disorders: an analysis of secondary measures. Biol Psychiatry. 2007 Feb 15;61(4):538-44. doi: 10.1016/j.biopsych.2006.09.028. PMID 17276750
- [Background] Sukhodolsky DG, Scahill L, Gadow KD, Arnold LE, Aman MG, McDougle CJ, McCracken JT, Tierney E, Williams White S, Lecavalier L, Vitiello B. Parent-rated anxiety symptoms in children with pervasive developmental disorders: frequency and association with core autism symptoms and cognitive functioning. J Abnorm Child Psychol. 2008 Jan;36(1):117-28. doi: 10.1007/s10802-007-9165-9. Epub 2007 Aug 3. PMID 17674186
- [Result] Research Units on Pediatric Psychopharmacology Autism Network. Randomized, controlled, crossover trial of methylphenidate in pervasive developmental disorders with hyperactivity. Arch Gen Psychiatry. 2005 Nov;62(11):1266-74. doi: 10.1001/archpsyc.62.11.1266. PMID 16275814
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- See also: More information on childhood disorders — http://www.nimh.nih.gov/health/topics/child-and-adolescent-mental-health/index.shtml